CLINICAL TRIAL: NCT04346134
Title: Miniaturized Percutaneous Nephrolithotomy Versus Extracorporeal Shock Wave Lithotripsy in Treatment of Non- Lower Polar, High-Density, Renal Stone of 10 to 20 mm Size: A Prospective, Randomized Study
Brief Title: Mini- Percutaneous Nephrolithotomy Versus Extracorporeal Shock Wave Lithotripsy for High Density Renal Stones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Abul-fotouh Ahmed, Professor of Urology and Andrology, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Uro_Azhar_16_019
Record Dates: First submitted 2020-04-13; First posted 2020-04-15 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-02

CONDITIONS: Renal Stone; Extracorporeal Shockwave Lithotripsy; Percutaneous Nephrolithotomy
MeSH Terms: conditions — Nephrolithiasis

STUDY DESIGN:
Intervention Model Description: Double-arm, prospective, Randomized, intervention study
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mini-PNL group (Experimental): In which percutaneous nephrolithotomy will be performed using miniature nephroscope.
  Interventions: Procedure: mini-PNL
- SWL group (Experimental): In which extracorporeal shock wave lithotripsy will be performed using Dornier lithotripter SII
  Interventions: Procedure: SWL

INTERVENTIONS:
Procedure: mini-PNL — Percutaneous nephrolithotomy using miniature nephroscope. The procedure will be performed under general or spinal anesthesia under fluoroscopy guidance.
  Arms: mini-PNL group
Procedure: SWL — Extracorporal shockwave lithotripsy using Dornier SII lithotripter. the procedure will be performed under sedoanalgesia, and fluoroscopy will be used for stone localization; for a maximum of 3 SWL session.
  Arms: SWL group

SUMMARY:
Several studies were conducted to compare extracorporeal shockwave lithotripsy (SWL) and percutaneous nephrolithotomy (PNL) as treatment options for medium size lower caliceal high dense stones. However, no studies compared these options for non- lower polar stones.

In the present study the investigators will compare mini-PNL and SWL in treatment of non- lower polar, medium size, high dense renal stones in reference to the stone free rate and safety of the procedures.

Pre-operative evaluation including abdominal non-contrasted computed tomography will be performed for all patients. Patients will be randomly allocated into two equal groups and will be treated by either mini-PNL or SWL. postoperative, patients will be followed by regularly for 3 months. the outcome of the procedures will be evaluated and compared between groups.

DETAILED DESCRIPTION:
The European guidelines put SWL and PNL as an equal treatment options for non- lower polar renal stones from 10 to 20 mm size regardless of density. However, several studies reported markedly reduced SFR after SWL with increased density. Also, in practice, the investigators noticed a high failure rate in renal stones with high density regardless of stone size. Several studies were conducted to compare SWL and PNL as treatment options for medium size lower caliceal stones. However, no studies compared these options for non- lower polar stones.

In the present study the investigators will compare mini-PNL and SWL in treatment of non- lower polar, medium size, high dense renal stones in reference to the SFR and safety of the procedures.

Adult patients with renal stones who agree to participate in the study will evaluated evaluated by full medical history taking and thorough physical examination, urinalysis, urine culture and antibiogram, complete blood cell count (CBC), serum creatinine, liver function tests and coagulation profile. Plain abdominal X-ray for kidney, ureters and urinary bladders (KUB), abdominal ultrasonography and abdominal non-contrasted computed tomography (NCCT). Preoperative assessment of renal anatomy and stone characteristics will be based on the findings of abdominal NCCT.

patients with high density (>1000 HU), non-lower polar, single renal stone of 10 to 20 mm size will be randomly divided into 2 equal groups. mini-PNL group, in which PNL procedures will be performed using miniature nephroscope and SWL group, in which SWL procedures will be performed using Dornier Lithotripter. SWL will be performed for a maximum of 3 sessions.

Patients will be followed up regularly, post-operatively for 3 months. NCCT will be performed after 3 months for detection of stone free status. Baseline data, intra-operative and post-operative parameters will be compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with high density (>1000 HU), non-lower polar, single renal stone of 10 to 20 mm size

Exclusion Criteria:

* Pregnant women, morbid obesity, severe orthopaedic deformities, any co-morbidities precluding general anaesthesia or prone positioning, uncorrectable coagulation disorders, active urinary tract infection (UTI), stone in calyceal diverticulum, abnormal renal anatomy and urinary tract obstruction distal to the stone

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2020-07-14 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Stone Free Rate | as detected by non-contrasted computed tomography 3 months after the intervention procedures.
  No residual renal stone or residual fragment(s) less than 4 mm size

SECONDARY OUTCOMES:
Complications | Intra- and 3 months post-operative complications

CONTACTS AND LOCATIONS:
Locations (1):
- Urology Department, Al-Azhar University Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided